CLINICAL TRIAL: NCT06549608
Title: Patient Characteristics and Treatment Duration of Mavacamten Obstructive HCM Patient Support Program in Canada: A Retrospective Cohort Study
Brief Title: A Retrospective Cohort Study of Mavacamten Patient Support Program in Canada
Status: Active, not recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV027-1187
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: Hypertrophic cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — MYK-461

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Adults participants treated with mavacamten: Participants with symptomatic obstructive hypertrophic cardiomyopathy (NYHA functional class II-III) who receive mavacamten as part of routine clinical care.
  Interventions: Drug: Mavacamten

INTERVENTIONS:
Drug: Mavacamten — As per product label

SUMMARY:
This real-world study will describe the demographic and clinical characteristics and mavacamten treatment of adult patients with obstructive hypertrophic cardiomyopathy who participated in the Bristol-Myers Squibb (BMS)-sponsored CAMZYOS Patient Support Program in Canada.

ELIGIBILITY:
Inclusion Criteria:

* Participants ≥18 years of age.
* Participants who have initiated mavacamten as part of routine clinical care, through the BMS-sponsored CAMZYOS Patient Support Program for the treatment of symptomatic obstructive hypertrophic cardiomyopathy.
* Participants who consented to the use of their de-identified data, generated from information collected in the course of the program.

Exclusion Criteria:

• There are no exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants in Canada diagnosed with hypertrophic cardiomyopathy (oHCM) receiving mavacamten treatment as part of the BMS-sponsored CAMZYOS Patient Support Program
Sampling Method: Non-Probability Sample
Enrollment: 685 (Actual)
Dates: Start 2024-04-20 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2025-04-18 (Estimated)

PRIMARY OUTCOMES:
Participant demographics | Baseline
Participant clinical characteristics | Baseline

SECONDARY OUTCOMES:
Dose regimen of mavacamten treatment | Every 3-months up to 14 months
Titration patterns of mavacamten treatment | Up to 14 months
Mavacamten treatment duration | Up to 14 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts